CLINICAL TRIAL: NCT01554280
Title: Fully, Coated, Removable, Self-expanding Oesophageal Stents for the Prevention of Oesophageal Stricture Following Endoscopic Mucosal Resection of Short Segment Barrett's With High Grade Dysplasia and Early Cancer.
Brief Title: Fully Coated, Removable, Self-expanding Oesophageal Stents for Preventing Strictures Following Complete Barretts Excision.
Acronym: CBE-001-SEOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Professor Michael Bourke (Other)
Responsible Party: Sponsor-Investigator, Professor Michael Bourke, Dr Michael Bourke, Western Sydney Local Health District
Organization: Western Sydney Local Health District (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CBE-001-SEOS
Record Dates: First submitted 2012-03-11; First posted 2012-03-14 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Constriction, Pathological
Keywords: Stricture; Dysphagia
MeSH Terms: conditions — Constriction, Pathologic; Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oesophageal Stents (Experimental): Patients enrolled will receive a fully coated, removable, self-expanding oesophageal stent.
  Interventions: Device: Fully coated, removable , self-expanding oesophageal stent

INTERVENTIONS:
Device: Fully coated, removable , self-expanding oesophageal stent — Insertion of the fully coated, removable, self-expanding oesophageal stent for the prevention of oesophageal strictures.

SUMMARY:
The purpose of this study is to investigate whether preventative placement of a removable oesophageal stent reduces the rate of scar tissue, or stricture formation after removing the precancerous or early cancerous Barrett's mucosa by Endoscopic Mucosal Resection (EMR). The stent will be placed 10-14 days after initial EMR. The stent will then be removed 8 weeks later by repeat Endoscopy. Patients will be followed up weekly following insertion of the oesophageal stent.

ELIGIBILITY:
Inclusion Criteria:

* Patients with short segment Barrett's Oesophagus with high grade dysplasia or early cancer, having circumferential EMR to achieve complete Barrett's excision.
* Aged 18-75 years old
* Biopsy proven to be Barretts with HGD or EAC
* The absence or lymph node involvement
* Short segment <3cm of Barretts Oesophagus.

Exclusion Criteria:

* Women who are pregnant and the human foetus
* Children and/or young people <18 years
* People with an intellectual or mental impairment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Improvement in Stricture Formation | 12 weeks
  Initial evaluation of Dysphagia score which is used to assess the stricture formation prior to EMR. Followed by weekly phone calls to assess ability to swallow liquids and food.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bourke, MBBS, Principal Investigator — WSLHD
Locations (1):
- Westmead Hospital, Westmead, New South Wales, Australia

REFERENCES:
- [Derived] Holt BA, Jayasekeran V, Williams SJ, Lee EY, Bahin FF, Sonson R, Lord RV, Bourke MJ. Early metal stent insertion fails to prevent stricturing after single-stage complete Barrett's excision for high-grade dysplasia and early cancer. Gastrointest Endosc. 2015 Apr;81(4):857-64. doi: 10.1016/j.gie.2014.08.022. Epub 2014 Oct 16. PMID 25442084